CLINICAL TRIAL: NCT00665964
Title: A Prospective, Randomized, Multi-center Study Comparing the Ten-Year Survival for X-3 Polyethylene to N2vac Polyethylene When Used With the Triathlon Posterior Stabilized (PS) Total Knee System
Brief Title: Comparing X-3 To N2vac Polyethylene With the Triathlon Total Knee System
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not funded at this time.
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Canada LP (Industry)
Responsible Party: Principal Investigator, Michael Dunbar, Principal Investigator, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA-RS/2007-249
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis; OA
Keywords: osteoarthritis; knee; total knee arthroplasty; gonarthrrsis; polyethylene; posterior stabilized
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- X-3 (Experimental): X-3 polyethylene which is a new highly cross-linked poly that is theorized to be more durable in vivo
  Interventions: Device: X-3 polyethylene
- N2Vac polethylene (Active Comparator): conventional polyethylene
  Interventions: Device: N2Vac polethylene

INTERVENTIONS:
Device: X-3 polyethylene — highly cross-linked polyethylene for knee arthroplasty
  Arms: X-3
Device: N2Vac polethylene — conventional polyethylene
  Arms: N2Vac polethylene

SUMMARY:
Methodology: This study will be a randomized, multi-center evaluation comparing N2vac polyethylene inserts and patellas with X3 inserts and patellas when used in the Triathlon PS total knee system.

Study Duration: 12-18 month enrollment period + 10 year follow-up for each case years total duration

Multi-centre study

Objectives

Primary: To compare the 10 year implant survival of the Triathlon PS total knee system when X3 polyethylene components are used to the same knee system when N2Vac components are used.

Secondary: To compare pain, function, radiographic outcomes, and health related quality of life of subjects in both treatment groups. Safety will be assessed by comparison of adverse events between the groups.

Number of Subjects 384 cases (197 each group)

ELIGIBILITY:
Inclusion Criteria:

* The subject requires a primary cemented total knee replacement.
* The subject has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
* The subject has intact collateral ligaments.
* The subject has signed the ethic committee approved, study specific Informed Patient Consent Form.
* The subject is willing and able to comply with post-operative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* The subject has inflammatory arthritis.
* The subject is morbidly obese, BMI > 40.
* The subject has a history of total or unicompartmental reconstruction of the affected joint.
* The subject has had a high tibial osteotomy or femoral osteotomy.
* The subject has a neuromuscular or neurosensory deficiency, that would limit the ability to assess the performance of the device.
* The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
* The subject is immunologically suppressed, or receiving chronic steroids (>30 days duration).
* The subject's bone stock is compromised by disease or infection and cannot provide adequate support and/or fixation to the prosthesis.
* The subject has had a knee fusion at the affected joint.
* The subject has an active or suspected latent infection in or about the knee joint.
* The subject is a prisoner.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
survival rate of polyethylene | 10 years

SECONDARY OUTCOMES:
pain | 10 years
function | 10 years
radiographic outcomes | 10 years
health related quality of life | 10 years
adverse events | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Dunbar, Principal Investigator — Dalhousie University
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada